CLINICAL TRIAL: NCT04896814
Title: Transcutaneous Tibial Nerve Stimulation as Treatment for Women With Primary Dysmenorrhea: A Randomized Controlled Trial
Brief Title: Transcutaneous Tibial Nerve Stimulation as Treatment for Women With Primary Dysmenorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, Marta Correyero-León, Doctorate student, University of Salamanca
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Tibial2021
Record Dates: First submitted 2021-05-09; First posted 2021-05-21 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Dysmenorrhea Primary
Keywords: Dysmenorrhea; Menstruation Disturbances
MeSH Terms: conditions — Dysmenorrhea; Menstruation Disturbances

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcutaneous tibial nerve stimulation (Experimental): The participant will receive an intervention session per week that will be held for a period of 12 weeks. The total application time will be 30 minutes. A symmetrical biphasic current will be applied, with a frequency of 20 Hz in continuous mode and a pulsed frequency of 200 µs.
  Interventions: Procedure: Transcutaneous tibial nerve stimulation
- Placebo (Placebo Comparator): The participant will receive one intervention session per week will be performed during a 12 weeks period time. The total application time will be 30 minutes. A discontinuous current at 2Hz frequency and a pulsed frequency of 50 µs, with 2 seconds of work and 10 seconds of pause will be applied in other localization.
  Interventions: Procedure: Placebo

INTERVENTIONS:
Procedure: Transcutaneous tibial nerve stimulation — The participant will be placed in the supine position with the soles of the feet together and the knees flexed and abducted at 90º. Two adhesive electrodes will be used for each leg. First one: 32 mm of diameter that will be placed in the posterior tibial nerve, that is, 4-5 cm cranial to the internal malleolus, between the posterior edge of the medial border of the tibia and the soleus tendon. Second one: 50x50 mm to be placed in the ipsilateral calcaneus. The electrodes will be connected to the NeuroTracTM PelviTone stimulation device. The stimulation range will be selected according to the tolerable pain limit for the patient, between 0.5 and 20 mA (adjustable in 1 mA levels).The intensity elevation will be allowed each time the patient perceives the fading of the previous sensation due to accommodation. Under no circumstances should the stimulation cause a painful feeling.
  Arms: Transcutaneous tibial nerve stimulation
Procedure: Placebo — The participant will be placed in the same position. Two 50 x 50 mm adhesive electrodes will be placed on the external face of the thigh, on a single leg. This area is outside the territory of the posterior tibial nerve. A discontinuous current at 2Hz frequency and a pulsed frequency of 50 µs, with 2 seconds of work and 10 seconds of pause will be applied. This simulated current being considered to be insufficient to achieve therapeutic effects in the body and to be outside of the usual ranges described in electrotherapy manuals regarding pain management. The intensity will be selected according to the paint limit level of the patient, between 0.5 and 60 mA (adjustable in 0.1 mA levels), where a low or moderate sensation of the patient will be sought, without muscle contraction.
  Arms: Placebo

SUMMARY:
The goal of this study is to verify whether transcutaneous stimulation of the posterior tibial nerve improves pain, quality of life and sleep deficiency in patients with pain related to their menstrual period in the short and medium-long term.

The hypothesis of the study states that by applying that method to the patients, a decrease or disappearance of pain in menstruation should happen, as well as an improvement in quality of life and sleep deficiency.

The study will consist of:

* An interview, lasting 30 minutes, in which the characteristics of the study will be explained. In case of wishing to participate, it will be required to sign the informed consent document and to fill out the medical history sheet.
* An evaluation phase: in which it will be necessary to fill out a number of questionnaires during two consecutive menstrual periods.
* An intervention phase: consisting of 12 30-minute treatment sessions, once a week. The patients will be randomly assigned to one of the two groups. In both groups, a current will be applied to different locations on the legs. The technique will be performed through four/two electrodes leg attached to the skin. This stimulation will not be painful at any time nor will it have harmful effects on the patients health. In this phase, the individual should continue filling out the questionnaires provided in each period. On the last day of treatment, a scale of satisfaction with the treatment will be retrieved.
* A re-evaluation phase: in which the individual shall fill out a number of questionnaires a month, 3 and 6 months after finishing the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 18 and 43.
* Women with regular menstrual cycles (range between 21 and 35 days).
* Women with a visual analogue scale (VAS) between 4 and 10 (moderate to severe pain) during at least 50% of annual menstrual cycles and / or during the last 3 cycles in the suprapubic area, abdomen, lower lumbar area , perineum and / or medial side of the thighs during the first and / or second day of your menstrual cycle.
* Sign the informed consent document to participate in the study.

Exclusion Criteria:

* Women on hormonal therapy or who have an Intrauterine Device implanted.
* Women diagnosed of secondary dysmenorrhea by their gynecologist (endometriosis, ovarian cyst, etc.) in the last 18 months.
* Women who have underwent a surgery during the study.
* Women who have underwent abdominal and pelvic surgery or who have given birth (vaginal or cesarean section) in the last 6 months.
* Women with lesions on the skin of the upper-internal face of the ankles (scars, erosions or cysts).
* Women who are pregnant or planning a pregnancy.
* Women with pacemakers, uncorrected coagulopathies, severe comorbid disorder, cancer (in the last 5 years or now), severe mental disorders or neuropathies that affect the nerves of the pelvis or lower extremities.
* Physiotherapy or electrotherapy treatments that are related to the pathology or study areas of the month prior to the start of the study.

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Changes in pain perception assessed using a 100 mm Visual Analogue Scale (VAS). | Once a month for 6 months. Thereafter, at 3 months and at 6 months.
  The scale will be self-administered. Minimum value 0. Maximum value 100. Higher score = Higher level of pain. Lower and lower scores mean a better result.
Changes in pain perception assessed using the Short-Form McGill Pain Questionnaire (SF-MPQ®). | Once a month for 6 months. Thereafter, at 3 months and at 6 months.
  The questionnaire will be self-administered. The total score ranges from 0 to 45. Higher score = Higher level of pain. Lower and lower scores mean a better result.
Changes in the non-steroidal anti-inflammatory drugs (NSAID) intake using a NSAID diary designed for this study. | Once a month for 6 months. Thereafter, at 3 months and at 6 months.
  The questionnaire will be self-administered.
Changes in life quality assessed using the SF36 Health Survey (SF-36v2®). | Once a month for 6 months. Thereafter, at 3 months and at 6 months.
  The questionnaire will be self-administered. Minimum value 0. Maximum value 100. The higher the score, the better the state of health.
Changes in sleep quality assessed using the Pittsburgh Sleep Quality Index (PSQI®). | Once a month for 6 months. Thereafter, at 3 months and at 6 months.
  The scale will be self-administered. The total score ranges from 0 to 21. The higher the score, the worse the sleep state.

SECONDARY OUTCOMES:
To assess the overall improvement and satisfaction of the treatment using the Patient Global Impression of Change (PGIC®) questionnaire. | At 5 months and at 11 months.
  The questionnaire will be self-administered. The total score ranges from 1 to 7. The higher the score, the worse the impression of change.
To assess the overall improvement and satisfaction of the treatment using a Likert Scale designed for this study. | At 5 months and at 11 months.
  The questionnaire will be self-administered. The scale qualitatively expresses the degree of agreement or disagreement with the treatment. The higher the score, the better the satisfaction with the treatment.
To collect the possible adverse reactions caused by the treatment. | Once a week for 12 weeks.
  It will be assessed using an adverse reactions questionnaire that was designed for the study. It will be self-administered. This questionnaire does not have minimum and maximum values, it is an open question.

CONTACTS AND LOCATIONS:
Overall Officials: Marta Correyero-León, Doc student, Principal Investigator — University of Salamanca; Inés Llamas-Ramos, PhD, Study Director — University of Salamanca
Locations (1):
- USalamanca, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: No